CLINICAL TRIAL: NCT06878326
Title: Resting-State Functional Connectivity as a Predictor of tDCS Effects in Adolescents With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Yvonne Han, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20250212003
Record Dates: First submitted 2025-03-11; First posted 2025-03-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder (ASD); Transcranial Direct Current Stimulation (tDCS); Electroencephalography
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cathodal active tDCS (Experimental): For cathodal tDCS condition, participants will receive cathodal stimulation on the dorsolateral prefrontal cortex with ramp up and ramp down mode for 10 seconds, eliciting a tingling sensation on the scalp that fades over seconds. Following that, a twenty-minute executive functional task will be initiated five minutes subsequent to the stimulation mode, and the stimulation will be terminated when the task ends.
  Interventions: Device: tDCS
- Anodal active tDCS (Experimental): For anodal tDCS condition, participants will receive anodal stimulation on the dorsolateral prefrontal cortex with ramp up and ramp down mode for 10 seconds, eliciting a tingling sensation on the scalp that fades over seconds. Following that, a twenty-minute executive functional task will be initiated five minutes subsequent to the stimulation mode, and the stimulation will be terminated when the task ends.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): For sham-tDCS condition, participants will receive initial stimulation with ramp up and ramp down mode for 30 seconds, eliciting a tingling sensation on the scalp then it will be discontinued. Participant will also receive the twenty-minute executive functional task five minutes subsequent to the stimulation mode.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Participant will receive three stimulation conditions: cathodal tDCS of the left DLPFC, anodal tDCS of the left DLPFC and sham-tDCS. The order of the conditions will be randomized and counterbalanced across participants, and the three stimulation conditions will be administered at least a week apart to avoid carry-over effects. The tDCS session will last for 20 minutes.

SUMMARY:
Background: Transcranial Direct Current Stimulation (tDCS) is a form of non-invasive brain stimulation that has aroused increased interests in the past decade. Not only that it is transient with little side-effects, and can be well-tolerated by children, it is also affordable and readily accessible, making it an appealing treatment option for autism spectrum disorder (ASD).

Objective: (1) To evaluate the therapeutic effects of tDCS on improving cognitive function in patients with ASD, (2) to better understand the neural mechanisms underlying the neuromodulation effects of tDCS in patients with ASD, and (3) to determine whether resting-state functional connectivity measures can predict the therapeutic effects of active tDCS in individuals with ASD.

Methods: To assess the therapeutic effects and neural mechanisms of tDCS, 90 adolescents with ASD (age 12-22 years) will receive three stimulation conditions: cathodal tDCS of the left DLPFC, anodal tDCS of the left DLPFC and sham-tDCS with at least a week apart each time. During the active tDCS or sham-tDCS condition, the participants will be administered a computerized test battery (Cambridge Neuropsychological Test Automated Battery, CANTAB®) to evaluate their cognitive function. EEG before and after the tDCS to evaluate the tDCS-induced alteration in their neural activity and functional connectivity.

Hypothesis: Drawing together the different evidence linking ASD with cortical hyper-excitability and disordered neural connectivity, as reviewed previously, the investigators hypothesize that, relative to a sham-tDCS condition, active cathodal (inhibitory) and anodal (excitatory) tDCS over the left DLPRC will induce stimulation-linked facilitation of learning and resultant improvement of cognitive functioning in patients with ASD.

In addition to the therapeutic effects of tDCS, enhanced neural connectivity, as indexed by altered level EEG theta coherence in patients with ASD, will mediate the beneficial effects of tDCS, relative to sham tDCS, on improvements in cognitive function. Moreover, resting-state functional connectivity will moderate the beneficial effects of active tDCS on cognitive function, relative to sham tDCS, such that participants with greater pre-treatment resting state functional connectively will evidence greater/less response to tDCS, relative to participants receiving sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* being 12-22 years old
* diagnosed with ASD given by registered psychiatrists or clinical psychologists according to the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) criteria of ASD
* able to communicate in Chinese

Exclusion Criteria:

* without a confirmed diagnosis from the clinical psychologist
* history of other neurological and psychiatric disorders and head trauma
* on psychiatric medication

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in CANTAB® cognitive test - Reaction Time (RTI) | During each stimulation session, last around 3mins
  RTI assesses motor and mental response speeds, reaction time, response accuracy and impulsivity. It consists of 30 trials with five potential targets and requires participants to make flexible responses as fast as possible to the target stimulus (shown in yellow). Specifically, movement and reaction time will be measured, where shorter duration reflects faster processing speed.
Change in CANTAB® cognitive test - Spatial Working Memory (SWM) | During each stimulation session, last around 6mins
  SWM assesses retention and manipulation of visuospatial information. The participant should find one yellow "token" in each of a number of boxes and use them to fill up an empty column on the right of the screen by selecting the boxes and using a process of elimination. Error selecting boxes that have already been found to be empty and revisiting boxes which have already been found to contain a token will be measured.
Change in CANTAB® cognitive test - Multitasking Test (MTT): Response Latencies | During each stimulation session, last around 8mins
  MTT assesses the ability to resolve the interference of task-irrelevant information (stroop-like effect). The test displays an arrow which can appear on either the left or right side of the screen and can point to either the left or right side. In each trial, participants are presented with a cue that indicates which button to press according to two different rules. And the rules that participants have to follow may change from trial to trial in a randomized order. Participant's response latencies will be measured.
Change in CANTAB® cognitive test - Multitasking Test (MTT): Error Scores | During each stimulation session, last around 8mins
  MTT assesses the ability to resolve the interference of task-irrelevant information (stroop-like effect). The test displays an arrow which can appear on either the left or right side of the screen and can point to either the left or right side. In each trial, participants are presented with a cue that indicates which button to press according to two different rules. And the rules that participants have to follow may change from trial to trial in a randomized order. Participant's error scores will be measured.
Changes in EEG theta coherence | Before tDCS session, Right after tDCS session (2 timepoints, up to 20 minutes)
  Each participant will be tested individually to collect EEG data. The participants' eyes-open resting condition will be assessed by EEG for 5 minutes, before and after the tDCS to evaluate the tDCS-induced alteration in their neural activity and functional connectivity. Raw data will be processed with the EEGLAB Toolbox using MATLAB® R2019a. Data from 19 electrodes will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Han, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong